CLINICAL TRIAL: NCT03399006
Title: Combined 3D Power Doppler Placental Volume and Vascular Flow Indices In the First Trimester of Pregnancy Could be a Specific Screening Toll in the Early Prediction Of Preeclampsia?.
Brief Title: Combined 3D Power Doppler Placental Volume and Vascular Flow Indices In the First Trimester of Pregnancy as Predictors Of Preeclampsia?.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 19
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia: women who developed preeclampsia. Preeclampsia was defined as a blood pressure 140/90 mmHg and proteinuria of 300 mg in 24 hours, or two readings of at least 2+ on dipstick analysis of midstream urine specimens if no 24-hour urine collection was available in absence of urinary tract infection
  Interventions: Device: 2D ultrasound; Device: Doppler Ultrasound; Device: 3D ultrasound
- Normal pregnancy: women with normal blood presure
  Interventions: Device: 2D ultrasound; Device: Doppler Ultrasound; Device: 3D ultrasound

INTERVENTIONS:
Device: 2D ultrasound — Trans-abdominal ultrasound examination was performed with the woman placed in a recumbent or semi recumbent position & carried out for measurement of fetal CRL and diagnosis of any major fetal defects
Device: Doppler Ultrasound — measurement of UtA-PI & UtA-RI. A sagittal section of the uterus was obtained For the Doppler studies, and the cervical canal and internal cervical os were identified. The transducer was gently tilted from side to side and color flow mapping was used to identify each UtA along the side of the cervix and uterus at the level of the internal os.
  When three similar consecutive waveforms had been obtained the UtA-PI and UtA-RI were measured, and the mean UtA-PI and UtA-RI of the left and right arteries were calculated.
Device: 3D ultrasound — 3D transabdominal ultrasound of the Placental volume: the transducer with a full bladder and the transducer placed perpendicular to the placenta to see the entire placenta. The adjustments to 3D placental scan were an angle of 70° and a maximum region of interest that allowed the full placental surface. The external limits of the placenta were defined by the basal plate and the chorionic plate excluding the myometrium. Another acquisition was done, if the quality criteria were not attained.
  After sonography, the placental volume was calculated with 4D View software (GE Healthcare) by a single operator. The calculation was done twice using the same image, and the time spent was recorded. The VOCAL mode with an angle of rotation of 30° was chosen; the axial plane was the reference; and the calipers were placed on either side of the placenta. With 6 planes, it was possible to reconstruct the volume measured in cubic centimeters.

SUMMARY:
200 women at risk factor for preeclampsia will be subjected to transabdominal Doppler ultrasonography for assessment of placental volume measurements, pulasatility index (PI) and resistivity index (RI) in both uterine arteries, and assessment of the placental volume and its vascular indices (VI, FI, VFI)

DETAILED DESCRIPTION:
Ultrasonography assessment: Woman underwent an abdominal ultrasonographic examination including color-Doppler techniques at the period of 11-14 weeks of gestations to assess the following data:

* Gestational age was determined from the onset of the last normal menstrual period; measurements of fetal crown-rump length (CRL) were done to confirm the fetal gestational age.
* The fetal viability and careful search for any fetal abnormalities present.
* The measurement of the pulsatility index (PI), the resistance index (RI) in the uterine arteries both on the left and right side, detection for the presence of notch and determine whether it is unilateral or bilateral.
* The time of examination was approximately 20 minutes.
* The ultrasound equipment used for both abdominal sonography and color Doppler technique was GE ultrasound machine (model?? ) equipped with pulsed and color Doppler options was used with the probe frequency of 7 MHz.

Trans-abdominal ultrasound examination was performed with the woman placed in a recumbent or semi recumbent position & carried out for measurement of fetal CRL and diagnosis of any major fetal defects and measurement of UtA-PI & UtA-RI. A sagittal section of the uterus was obtained For the Doppler studies, and the cervical canal and internal cervical os were identified. The transducer was gently tilted from side to side and color flow mapping was used to identify each UtA along the side of the cervix and uterus at the level of the internal os.

the sampling gate set at 2mm to cover the whole vessel and care was taken to ensure that the angle of insonation was less than 60◦. When three similar consecutive waveforms had been obtained the UtA-PI and UtA-RI were measured, and the mean UtA-PI and UtA-RI of the left and right arteries were calculated.

Uterine artery Doppler was obtained with the patient in a semirecumbent position following a previously described technique [14]. A sagittal view of the uterus and of the cervical canal was obtained and color flow mapping was used to identify the uterine arteries coursing along the side of the cervix and uterus. The pulsed Doppler sample volume was placed on the ascending branch of the uterine artery closest to the internal os. The pulsatility index (PI = S _ D/M) was measured on three consecutive waveforms and the mean value between the left and right arteries was calculated. The presence of an early diastolic notch in the waveforms was recorded. An abnormal value was considered a mean PI greater than 2.36 corresponding to the 95th centile of a cross-sectional study on 3045 pregnancies

3D transabdominal ultrasound of the Placental volume: the transducer with a full bladder and the transducer placed perpendicular to the placenta to see the entire placenta. The adjustments to 3D placental scan were an angle of 70° and a maximum region of interest that allowed the full placental surface. The external limits of the placenta were defined by the basal plate and the chorionic plate excluding the myometrium. Another acquisition was done, if the quality criteria were not attained.

After sonography, the placental volume was calculated with 4D View software (GE Healthcare) by a single operator. The calculation was done twice using the same image, and the time spent was recorded. The VOCAL mode with an angle of rotation of 30° was chosen; the axial plane was the reference; and the calipers were placed on either side of the placenta. With 6 planes, it was possible to reconstruct the volume measured in cubic centimeters

ELIGIBILITY:
Inclusion Criteria:

* 1. Singleton pregnancy. 2. Familial history of preeclampsia as it has agenetic predisposition. 3. Regular menstrual cycles before pregnancy. 4. Females had preeclampsia in a previous pregnancy. 5. Gestational diabetes or essential hypertension or chronic nephritis with pregnancy" they will be seen between 11 - 14 weeks' of gestation

Exclusion Criteria:

* 1. Cases with fetal anomalies. 2. Dead fetuses

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: women at risk factor of preeclampsia as women with singleton pregnancy especially at the extremes of reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Development of preeclampsia | 28 to 38 weeks of gestational age
  Preeclampsia was defined as a blood pressure 140/90 mmHg and proteinuria of 300 mg in 24 hours, or two readings of at least 2+ on dipstick analysis of midstream urine specimens if no 24-hour urine collection was available in absence of urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided